CLINICAL TRIAL: NCT04646707
Title: Effect of Erector Spinae (ESP) Block on Opioid Reduction and Enhanced Recovery After Posterior Cervical Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-5818
Record Dates: First submitted 2019-11-05; First posted 2020-11-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Postoperative; Pain
Keywords: Opioid; Reduction; Enhanced; Postoperative; Recovery
MeSH Terms: conditions — Pain | interventions — Parapsychology; Dental Occlusion; Lidocaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: This is a double blind, randomized control clinical trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Bilateral ESP block at T1 level with 20 ml of 1:1 mixture (2% Lidocaine: 0.5% bupivacaine)
  Interventions: Drug: Erector Spinae (ESP) Block with Lidocaine/Bupivacaine
- Placebo Group (Placebo Comparator): Bilateral ESP block at T1 level with 20 ml of 0.9% normal saline
  Interventions: Drug: Erector Spinae (ESP) Block with placebo

INTERVENTIONS:
Drug: Erector Spinae (ESP) Block with Lidocaine/Bupivacaine — Bilateral ESP block at T1 level with 20 ml of 1:1 mixture (2% Lidocaine: 0.5% bupivacaine)
  Other Names: Study group
  Arms: Study group
Drug: Erector Spinae (ESP) Block with placebo — Bilateral ESP block at T1 level with 20 ml of 0.9% normal saline
  Other Names: Placebo group
  Arms: Placebo Group

SUMMARY:
Patients undergoing spine surgery frequently experience significant pain after surgery. This can limit patient activity and hinder rehabilitation. If inadequately treated, severe pain can result in emotional and psychological distress and ultimately impact long-term function, and increase the risk of developing pain that lasts longer than six months associated with depression, anxiety and disability.

More specifically, Erector Spinae Plane (ESP) block is a recently described plane block designed to block the dorsal and ventral rami of the thoracic spinal nerves. It has shown to be an effective modality for postoperative pain management as a part of multimodal analgesia in spinal surgery.

DETAILED DESCRIPTION:
Patients undergoing spine surgery frequently experience significant pain after surgery. Currently, standard management of acute pain after surgery consists mainly of systemic opioid narcotics and nonsteroidal anti-inflammatory drugs (NSAIDs). Generally, opiates and NSAIDs are not completely effective at managing pain, and they carry significant risk of addiction and overdose, particularly with prolonged or increased dosing. The concept of multimodal or ''balanced'' analgesia is rapidly becoming the 'standard of care' for preventing post-operative pain. It consists of the use of combinations of analgesics of different classes with different sites of action in an attempt to provide superior pain relief with reduced analgesic related side effects. Local anesthetic injection to block specific nerves has been widely recognized as a useful adjunct in a multimodal approach to postoperative pain management.

Erector Spinae Plane (ESP) block is a recently described plane block designed to block the dorsal and ventral rami of the thoracic spinal nerves. It has shown to be an effective modality for postoperative pain management as a part of multimodal analgesia in spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

All adult patients aged 18-80 years with ASA class I - III undergoing posterior cervical (C3-T2) decompression and instrumented fusion for cervical stenosis in prone position.

Exclusion Criteria:

1. In patients who are allergic to local anesthetics.
2. ASA IV patients
3. Lack of informed consent
4. Pregnant patient.
5. Fracture cervical spine
6. Extradural or intradural cervical tumors
7. Surgery of C1 and C2 spine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2025-12-17 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery 40 Questionnaire | 24 hours after surgery.
  the global Quality of Recovery-40 aggregate score is a scale from (1 to 5, where: 1 = very poor and 5 = excellent)

SECONDARY OUTCOMES:
Postoperative pain | 2 weeks and one month
  is a visual analog scale from (1 to 10, where: 1 is the mildest and 10 the worst possible)
Opioids consumption | 2 weeks and one month
  Patient Opioid/Non-Opioid Pain Medications Diary Card After Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dinsmore, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital?UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No